CLINICAL TRIAL: NCT00297791
Title: A Randomized Clinical Trial Comparing Laparoscopic and Open Surgery for Rectal Cancer.
Brief Title: COLOR II: Laparoscopic Versus Open Rectal Cancer Removal
Acronym: COLORII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDHA007
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2013-07

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; laparoscopic technique; open technique; clinical trial; multicenter study; randomized controlled trial; Tumor Below 15cm; curative surgical resection; no evidence for distant metastases
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): surgery (open or laparoscopic) and observation
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — randomized to open or laparoscopic technique
  Other Names: observation following intervention

SUMMARY:
COLOR II is a randomized, international, multi center study comparing the outcomes of laparoscopic and conventional resection of rectal carcinoma below 15 cm with curative intent. Clinical and operative data will be collected centrally in the coordinating centre in Halifax, Canada. Quality of life and costs will be assessed on a national basis.

DETAILED DESCRIPTION:
The design involves allocation of all suitable consecutive patients with rectal carcinoma to either of the two procedures at a randomization ratio of 2:1 in favor of the laparoscopic procedure. Excluded are patients with a carcinoma treated by local resection and palliative resections. The trial will be stratified according to participating centre, resection type, and preoperative radiotherapy.

If the 95% CI for the difference of the 3-year locoregional recurrence rates excludes a difference greater than 5% in favor of the conventional procedure, non-inferiority of the laparoscopic procedure will be concluded. Assuming both rates are 10%, 1000 evaluable cases are required in total for a power of 80%.

Analysis will be primarily on an intention to treat basis. Definition of conversion is defined by protocol.

ELIGIBILITY:
Inclusion Criteria:

* solitary rectal cancer observed at colonoscopy or on barium X-ray
* no evidence of distant metastases
* distal border of the tumor within 15 cm of the anal verge at rigid rectoscopy or under linea conjugata at lateral barium enema radiography
* suitable for elective surgical resection
* informed consent

Exclusion Criteria:

* T1 tumors treated by locl excision
* T4 tumors
* patients under 18 years of age
* signs of acute intestinal obstruction
* more than one colorectal tumor
* Familial Adenomatosis Polyposis, Hereditary Non-Polyposis Colorectal Cancer
* active crohn's or active ulcerative colitis
* scheduled need for other synchronous colon surgery
* preoperative indication of invasion of adjacent organs, immobile at palpation or CT showing invasion
* preoperative evidence of metastases (at least chest X-ray and liver ultrasound)
* other malignancies in medical history except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri
* absolute contraindications to general anesthesia or prolonged pneumoperitoneum (ASA class > III)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2004-06; Primary Completion 2013-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
locoregional recurrence rate | 3 years post operatively

SECONDARY OUTCOMES:
survival free of cancer recurrence | three, five and seven years post-operatively
overall survival | three, five and seven years post-operatively
port-site and wound-site recurrences | annually for seven years
distant metastases rate | annually for seven years
operative mortality and morbidity | 8 week or in-hospital
macroscopic evaluation of the resected specimen | post-operative
duration of in-hospital stay | post-operative
duration of absence of work | 8 weeks and 6 months post-operatively
postoperative health related quality of life,including standardized questionnaires on sexual and bladder function | weekly for 8 weeks
in-hospital direct and indirect costs | seven years
out-of-hospital postoperative costs | seven years

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Bonjer, MD, PhD, Principal Investigator — Dalhousie University, and VUMC, the Netherlands; Marius Hoogerboord, Principal Investigator — Nova Scotia Health Authority
Locations (35):
- Universitair Ziekenjuis Leuven, Leuven, Belgium
- Canada (3):
  - Royal Alexandra Hospital, University of Alberta, Edmonton, Alberta
  - CDHA/ Dalhousie University, Halifax, Nova Scotia
  - University of Western Ontario, London, Ontario
- Denmark (7):
  - Aalborg Hospital, Aalborg
  - SVS Esbjerg, Esbjerg
  - Amtssygehus i Gentofte, Gentofte Municipality
  - Hilleröd Hospital, Hilleröd
  - Odense Universitetshospital, Odense
  - Roskilde Hospital, Roskilde
  - Viborg, Viborg
- Germany (5):
  - Ludwig-Maximilians Universität Klinikum Großhadern, München
  - Caritas-Krankenhaus St. Josef, Regensburg
  - University Hospital Regensburg, Regensburg
  - Marienhospital, Stuttgart
  - Wuerzburg University, Würzburg
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Academisch Medisch Centrum, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - VU Medisch Centrum, Amsterdam
  - Rijnland Ziekenhuis, Leiderdorp
  - Erasmus Medical Centre, Rotterdam
  - Medisch Centrum Rijnmond-Zuid, Rotterdam
- Jagiellonian University, Krakow, Poland
- Korea University Anam Hospital, Seoul, South Korea
- Spain (5):
  - Hospital Clinic i Provencial de Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital S.A.S. de Jerez, Cadiz
  - Hospital del Sureste de Madrid, Madrid
  - Arrixaca Hospital Universitario, Murcia
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Örebro Hospital, Örebro
  - Kärnsjukhuset, Skvöde
  - Ersta Hospital, Stockholm
  - Uddevalla Hospital, Uddevalla

REFERENCES:
- [Derived] Andersson J, Angenete E, Gellerstedt M, Haglind E. Developing a multivariable prediction model of global health-related quality of life in patients treated for rectal cancer: a prospective study in five countries. Int J Colorectal Dis. 2024 Mar 5;39(1):35. doi: 10.1007/s00384-024-04605-y. PMID 38441657
- [Derived] Koedam TWA, Bootsma BT, Deijen CL, van de Brug T, Kazemier G, Cuesta MA, Furst A, Lacy AM, Haglind E, Tuynman JB, Daams F, Bonjer HJ; on behalf of the COLOR COLOR II study group. Oncological Outcomes After Anastomotic Leakage After Surgery for Colon or Rectal Cancer: Increased Risk of Local Recurrence. Ann Surg. 2022 Feb 1;275(2):e420-e427. doi: 10.1097/SLA.0000000000003889. PMID 32224742
- [Derived] Petersson J, Koedam TW, Bonjer HJ, Andersson J, Angenete E, Bock D, Cuesta MA, Deijen CL, Furst A, Lacy AM, Rosenberg J, Haglind E; COlorectal cancer Laparoscopic or Open Resection (COLOR) II Study Group. Bowel Obstruction and Ventral Hernia After Laparoscopic Versus Open Surgery for Rectal Cancer in A Randomized Trial (COLOR II). Ann Surg. 2019 Jan;269(1):53-57. doi: 10.1097/SLA.0000000000002790. PMID 29746337
- [Derived] Bonjer HJ, Deijen CL, Abis GA, Cuesta MA, van der Pas MH, de Lange-de Klerk ES, Lacy AM, Bemelman WA, Andersson J, Angenete E, Rosenberg J, Fuerst A, Haglind E; COLOR II Study Group. A randomized trial of laparoscopic versus open surgery for rectal cancer. N Engl J Med. 2015 Apr 2;372(14):1324-32. doi: 10.1056/NEJMoa1414882. PMID 25830422
- [Derived] Andersson J, Abis G, Gellerstedt M, Angenete E, Angeras U, Cuesta MA, Jess P, Rosenberg J, Bonjer HJ, Haglind E. Patient-reported genitourinary dysfunction after laparoscopic and open rectal cancer surgery in a randomized trial (COLOR II). Br J Surg. 2014 Sep;101(10):1272-9. doi: 10.1002/bjs.9550. Epub 2014 Jun 12. PMID 24924798
- [Derived] Andersson J, Angenete E, Gellerstedt M, Angeras U, Jess P, Rosenberg J, Furst A, Bonjer J, Haglind E. Health-related quality of life after laparoscopic and open surgery for rectal cancer in a randomized trial. Br J Surg. 2013 Jun;100(7):941-9. doi: 10.1002/bjs.9144. PMID 23640671
- [Derived] van der Pas MH, Haglind E, Cuesta MA, Furst A, Lacy AM, Hop WC, Bonjer HJ; COlorectal cancer Laparoscopic or Open Resection II (COLOR II) Study Group. Laparoscopic versus open surgery for rectal cancer (COLOR II): short-term outcomes of a randomised, phase 3 trial. Lancet Oncol. 2013 Mar;14(3):210-8. doi: 10.1016/S1470-2045(13)70016-0. Epub 2013 Feb 6. PMID 23395398
- [Derived] Color II Study Group; Buunen M, Bonjer HJ, Hop WC, Haglind E, Kurlberg G, Rosenberg J, Lacy AM, Cuesta MA, D'Hoore A, Furst A, Lange JF, Jess P, Bulut O, Poornoroozy P, Jensen KJ, Christensen MM, Lundhus E, Ovesen H, Birch D, Iesalnieks I, Jager C, Kreis M, van riet Y, van der Harst E, Gerhards MF, Bemelman WA, Hansson BM, Neijenhuis PA, Prins HA, Balague C, Targarona E, Lujan Mompean JA, Franco Osorio JD, Garcia Molina FJ, Skullman S, Lackberg Z, Kressner U, Matthiessen P, Kim SH, Poza AA. COLOR II. A randomized clinical trial comparing laparoscopic and open surgery for rectal cancer. Dan Med Bull. 2009 May;56(2):89-91. PMID 19486621